CLINICAL TRIAL: NCT01220336
Title: Study of Medical Assistant Health Coaching in Primary Care for Patients With Chronic Conditions
Acronym: HCPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ellen Chen, Adjunct Faculty, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UCSF CEPC
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Coaching (Experimental)
  Interventions: Behavioral: Health coaching by medical assistants in primary care

INTERVENTIONS:
Behavioral: Health coaching by medical assistants in primary care — Patients with uncontrolled diabetes, hypertension, hyperlipidemia will receive health coaching by medical assistants working with primary care providers in the Teamlet Model [Bodenheimer 2007] for 12 months.

SUMMARY:
Randomized control trial studying the effect of medical assistant health coaching for patients with diabetes, hypertension and hyperlipidemia within two San Francisco primary care community clinics, Mission Neighborhood Health Center and Southeast Health Center

ELIGIBILITY:
Inclusion Criteria:

Active patients at Mission Neighborhood Health Center, SF, USA or Southeast Health Center, SF, USA age 18-75 years Uncontrolled diabetes II, hypertension or hyperlipidemia Spanish or English speaking

Exclusion Criteria:

Cognitive dysfunction, mental health or physical condition that prevents participation in health coaching.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Composite clinical outcome measure- improvement in either HgA1C, SBP, or LDL | 12 months

SECONDARY OUTCOMES:
Composite clinical outcome measure- improvement in either HgA1C, SBP, or LDL | 24 months
  This second measurement of clinical outcomes will occurs one year after the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Chen, MD, Principal Investigator — University of California, San Francisco; David Thom, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Mission Neighborhood Health Center, San Francisco, California
  - Southeast Health Center, San Francisco, California

REFERENCES:
- [Derived] Willard-Grace R, DeVore D, Chen EH, Hessler D, Bodenheimer T, Thom DH. The effectiveness of medical assistant health coaching for low-income patients with uncontrolled diabetes, hypertension, and hyperlipidemia: protocol for a randomized controlled trial and baseline characteristics of the study population. BMC Fam Pract. 2013 Feb 23;14:27. doi: 10.1186/1471-2296-14-27. PMID 23433349